CLINICAL TRIAL: NCT06445959
Title: Phase 1b/2 Study of Decitabine and Venetoclax in Combination With the Targeted Mutant IDH1 Inhibitor Olutasidenib
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Rigel Pharmaceuticals,Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0180; NCI-2024-04807 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Mutant IDH1 Inhibitor Olutasidenib
MeSH Terms: interventions — olutasidenib; venetoclax; Decitabine; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Participants enrolled in Part 1, the dose of venetoclax/decitabine you receive will depend on when you join this study. Up to 3 dose levels will be tested. Up to 6 participants will be enrolled at each dose level.
  - All participants will receive the same dose level of olutasidenib.
  Interventions: Drug: Olutasidenib; Drug: Venetoclax; Drug: Decitabine; Drug: Decitabine/cedazuridine
- Part 2 (Experimental): Participants enrolled in Part 2, you will receive venetoclax/decitabine at the recommended dose that was found in Part 1.
  - All participants will receive the same dose level of olutasidenib.
  Interventions: Drug: Olutasidenib; Drug: Venetoclax; Drug: Decitabine; Drug: Decitabine/cedazuridine

INTERVENTIONS:
Drug: Olutasidenib — Given by PO
Drug: Venetoclax — Given by PO
  Other Names: ABT-199; GDC-0199
Drug: Decitabine — Given by IV
  Other Names: Dacogen
Drug: Decitabine/cedazuridine — Given by PO
  Other Names: INQOVI; ASTX727

SUMMARY:
To find a recommended combination dose of decitabine and venetoclax that can be given in combination with olutasidenib to participants with AML.

DETAILED DESCRIPTION:
Primary Objectives

* Phase 1b: To determine the safety and tolerability and recommended phase 2 dose (RP2D) of decitabine (either IV or oral decitabine/cedazuridine (ASTX727, Inqovi)) and venetoclax in combination with olutasidenib.
* Phase 2: To determine the composite remission rate (CR, CRh and CRi) of decitabine (IV or oral decitabine/cedazuridine (ASTX727, Inqovi)) and venetoclax in combination with olutasidenib for newly diagnosed (Arm A) or relapsed/refractory (Arm B) participants with IDH1-mutated myeloid malignancy.

Secondary Objectives

* To determine duration of response (DOR), event-free survival (EFS), and overall survival (OS)
* To evaluate occurrence of minimal residual disease (MRD) negative status by multiparameter flow cytometry and molecular evaluation.
* To determine the overall response rate (CR, CRh, CRi, MLFS, and PR)
* To characterize the pharmacokinetic (PK) profiles of venetoclax and olutasidenib in plasma samples (Phase 1b only).

Exploratory Objectives

- To investigate global gene expression profiles, DNA methylation profiles, BH3 profiling and other potential prognostic markers to explore predictors of antitumor activity and/or resistance to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Participants must have a documented IDH1 gene mutation
3. Participants with a diagnosis of relapsed or refractory AML (including biphenotypic or bilineage leukemia including a myeloid component or isolated extramedullary AML), high-risk MDS by IPSS-R or IPSS-M; OR
4. Participants with newly diagnosed AML not eligible or appropriate for intensive chemotherapy are also eligible. (Phase 2 portion only)
5. To be considered not eligible for intensive chemotherapy, participants must be defined by the following: Age 75 years or older, or Age 18 to 74 years with at least one of the following comorbidities:

   1. Severe cardiac disorder (eg, congestive heart failure requiring treatment, ejection fraction ≤50%, or chronic stable angina).
   2. Severe pulmonary disorder (eg, DLCO ≤65% or forced expiratory volume in 1 second [FEV1] ≤65%).
   3. Creatinine clearance ≥30 mL/min to <45 mL/min.
   4. Moderate hepatic impairment with total bilirubin >1.5 to .3.0 x upper limit of normal (ULN)
   5. ECOG performance status of 2 or 3
   6. Any other comorbidity that per the investigator renders a patient inappropriate for intensive chemotherapy
6. Eastern Cooperative Oncology Group (ECOG) Performance Status </=2 (unless age 18 to 74 years of age with newly diagnosed AML not eligible for intensive chemotherapy as per 5e above)
7. Adequate renal function including creatinine < 1.5, unless related to the disease or unless age 18 to 74 years of age with newly diagnosed AML not eligible for intensive chemotherapy as per 5c above.
8. Adequate hepatic function (direct bilirubin < 2x upper limit of normal (ULN) unless increase is due to Gilbert fs disease or leukemic involvement, and AST and/or ALT < 3x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT < 5x ULN will be considered eligible, or unless age 18 to 74 years of age with newly diagnosed AML not eligible for intensive chemotherapy as per 5d above)
9. In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 14 days for cytotoxic or non-cytotoxic (immunotherapy agent(s), or an interval of 5 half-lives of the prior therapy. Oral hydroxyurea and/or cytarabine (up to 2 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the PI. Concurrent intrathecal therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted.
10. Male participants who are sexually active with a women of childbearing potential (WOCBP) and who have not had vasectomies must be willing to use a barrier method of contraception and refrain from sperm donation from initial study drug until 90 days after last dose of study drug.
11. Willing and able to provide informed consent.

Exclusion Criteria:

1. Participants with t(15;17) karyotypic abnormality or acute promyelocytic leukemia (French-American-British [FAB] class M3-AML).
2. Participants with any concurrent uncontrolled clinically significant medical condition including life-threatening severe infection, or psychiatric illness, which could place the participants at unacceptable risk of study treatment.
3. Participants with active, uncontrolled leukemia involvement of the CNS
4. Participants with active graft-versus-host-disease (GVHD) status post stem cell transplant including active cGVHD requiring topic therapy. Patients must have discontinued calcineurin inhibitors at least 4 weeks prior to start of study treatment.
5. Participants with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
6. Known active hepatitis B (HBV) or Hepatitis C (HCV) infection or known HIV infection.
7. Participant has a white blood cell count > 25 x 10^9/L. (Note: Hydroxyurea and cytarabine is permitted to meet this criterion.)
8. Nursing women, women of childbearing potential (WOCBP) with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception.

A) Appropriate highly effective method(s) of contraception include oral or injectable hormonal birth control, IUD, and double barrier methods (for example a condom in combination with a spermicide).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org